CLINICAL TRIAL: NCT00840320
Title: A Phase I, Randomized, Single-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Repeat Oral Doses of 1278863A in Healthy Subjects
Brief Title: Repeat Dose Safety Study for Compound to Treat Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 112842
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Kidney Disease
Keywords: Safety; tolerability
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Repeat doses of active at escalating doses
  Interventions: Drug: 1278863
- 2 (Placebo Comparator): Repeat doses of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1278863 — 15mg, 25mg, 50mg, 150mg
  Arms: 1
Drug: Placebo — matching placebo
  Arms: 2

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of repeat doses of compound 1278863A in healthy subjects.

DETAILED DESCRIPTION:
Compound 1278863A is a novel small molecule agent, which stimulates erythropoiesis through inhibition of hypoxia-inducible factor (HIF)-prolyl hydroxylases (EGLNs). This compound is being developed for the treatment of anemia. Compound 111427 was the first administration of compound 1278863A to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single oral doses up to 300 mg in healthy adult subjects. This study, PHI112842, will be the first administration of compound 1278863A to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of repeat oral doses up to 300 mg for 14 days in healthy adult subjects. At least 6 subjects will complete each cohort. Multiple blood samples for pharmacokinetic analyses will be obtained post-dose in each cohort. Safety will be assessed by measurement of vital signs, cardiac monitoring, collection of adverse event assessments and laboratory safety tests. Blood samples will be collected for pharmacodynamic analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
2. Male or female between 18 and 55 years of age, inclusive.
3. A female subject must be of non-childbearing potential.
4. Male subjects must agree to use one of the acceptable contraception methods listed in the protocol
5. Body weight greater than or equal to 50 kg and BMI within the range 19 - 31 kg/m2 (inclusive).
6. Capable of giving written informed consent
7. QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

1. The subject has a positive pre-study drug screen.
2. A hemoglobin value at screening is:

   * Male subjects or post-menopausal females: > 15.5 g/dL
   * Female subjects: > 14.5 g/dL
3. The values of hematological parameters at screening are:

   MCV: outside the reference range and clinically significant deemed by the investigator and GSK Medical Monitor
4. The values of the following tests at screening are:

   * TIBC: outside the reference range
   * Serum iron: outside the reference range
   * Serum ferritin: outside the reference range
5. A value at screening is greater than the upper limit of reference range for the following clinical laboratory parameters: AST, ALT, direct bilirubin.
6. Clinically significant abnormal CPK determined by the investigator and GSK Medical Monitor.
7. Calculated creatinine clearance: < 60mL/min
8. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
9. A positive test for HIV antibody.
10. History of drug abuse or dependence within 6 months of the study.
11. History of regular alcohol consumption within 6 months of the study
12. Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
13. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study drug
14. History of sensitivity to any of the study drugs, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
15. History of sensitivity to heparin or heparin-induced thrombocytopenia. (if the clinical research unit uses heparin to maintain intravenous cannula patency)
16. Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, and/or hepatic function that could interfere with the absorption, metabolism, and/or excretion of the study drugs.
17. History of peptic ulcer disease.
18. History of malignancy tumor. Non-melanoma skin cancer that has been definitely removed is allowed.
19. Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
20. Lactating females.
21. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
22. Unwillingness or inability to follow the procedures, or lifestyle and/or dietary restrictions outlined in the protocol.
23. Consumption of red wine, seville oranges, grapefruit or grapefruit juice, exotic citrus fruits, grapefruit hybrids or fruit juices of the prohibited fruits from 7 days prior to the first dose of study medication
24. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
25. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
26. Subject is mentally or legally incapacitated.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-03-13 (Actual); Primary Completion 2009-09-02 (Actual); Study Completion 2009-09-02 (Actual)

PRIMARY OUTCOMES:
adverse events reporting | throughout study
Safety Labs (hematology) | Screening, Days -1, 1-3, 5, 7, 9, 11, 14-18, 21, 25, 28
vital signs (blood pressure and heart rate) | Days 1-15, 28
12-lead ECG | Screening, Days 1-2, 4, 6, 8, 10, 12, 14, 28
dual-lead cardiac monitoring (telemetry monitoring) | Days -1 to 3, 14
clinical monitoring/observation | throughout
Safety Labs (Chemistry) | Screening, Days -1, 1-3, 7, 10, 14-15, 17, 21, 28
Safety Labs (Urinalysis) | Screening, Days -1, 1-3, 7, 10, 14-15, 17, 21, 28

SECONDARY OUTCOMES:
AUC(0-∞) on Day 1, AUC(0-τ), Cmax, tmax and t1/2, on Days 1 and 14 | Days 1-2, 4, 6, 8, 10, 12, 14-18
Trough plasma concentrations at the end of the dosing interval | Days 2, 4, 6, 8, 10 and 12
Hemoglobin actual values, rate of rise, maximum change from baseline, and rate of decline following stopping of dosing | Days 1, 7, 14, 21, 28
Fetal hemoglobin actual values, change from baseline, and percent of total hemoglobin | Days 1, 7, 14, 21, 28
Actual values and change from baseline in erythropoietin | Days 1-4, 7, 14-15, 18, 21
Actual values and change from baseline in absolute VEGF | Days 1-2, 14-15, 18, 21
Actual values and change from baseline in hepcidin | Days 1-2, 7, 14-15, 18, 21
Actual values and change from baseline in total iron binding capacity (TIBC) | Screening, Days 1, 7, 14, 18, 21
Actual values and change from baseline in transferring saturation (%) | Days 1, 7, 14, 18, 21

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Melbourne, Victoria, Australia

REFERENCES:
- See also: Results for study 112842 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112842?search=study&search_terms=112842#rs